CLINICAL TRIAL: NCT04804124
Title: Sleep Duration and Cardiovascular Health
Acronym: Goldilocks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Saurabh Thosar, Assistant Professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00021448
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Sleep; Cardiovascular Risk Factor
Keywords: cardiovascular; sleep duration; vascular endothelial function

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Sleepers (Experimental): Reported nightly sleep time of ≤6 hours
  Interventions: Behavioral: Regularized Sleep Schedule
- Long Sleepers (Experimental): Reported nightly sleep time of ≥9 hours
  Interventions: Behavioral: Regularized Sleep Schedule
- Average Duration Sleepers (Experimental): Reported nightly sleep time of 7-8 hours
  Interventions: Behavioral: Regularized Sleep Schedule

INTERVENTIONS:
Behavioral: Regularized Sleep Schedule — Participants may maintain a self-selected 8-hour per night sleep schedule as an optional intervention. Participants from any of the three groups may complete the intervention.

SUMMARY:
This is a cross-sectional study with an optional intervention that will examine how extreme sleep durations relate to cardiovascular health, physical activity, and sleep quality by studying three groups of participants: short sleepers (≤ 6 hrs), long sleepers (≥ 9 hrs), and average duration sleepers (7-8 hrs). The optional intervention asks participants to maintain an 8-hour per night regular sleep schedule for one week.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To test the hypothesis that vascular endothelial function in the brachial artery, and other associated cardiovascular risk markers are impaired in short sleepers and long sleepers as compared to the control group of average duration sleepers.

To test the hypothesis that the optional intervention to maintain an 8-hour per night sleep schedule will alleviate vascular endothelial function impairment.

OUTLINE:

Participants will measure sleep, physical activity, and blood pressure with at-home devices before coming in for one in-lab visit, where they will have vascular function and blood markers measured, as well as an optional CT scan to measure calcium in the coronary arteries. An optional intervention may occur after this: Participants will continue the at-home measures while maintaining a chosen regular 8-hour per night sleep schedule, before coming in for a second in-lab visit with all same measures except for CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 25-65y
* Lean and overweight (BMI 18.5-40 kg/m2)
* No acute, chronic, or debilitating medical conditions
* No prescription/non-prescription medications or drugs of abuse
* Current non-smoker (tobacco and marijuana)
* Persons who fit all the above criteria and are suitable based on a medical history and health habits questionnaire, and additional sleep and health profiling questionnaires may be eligible to participate.

Exclusion Criteria:

* Persons with any acute, chronic, or debilitating medical condition except pre-hypertension will be excluded.
* Persons with any symptoms of acute or active illness (e.g. fever, leukocytosis) will be excluded.
* Persons with a history of severe psychiatric illness or psychiatric disorders will be excluded.
* Persons with a history of regular night/or rotating shift work in the past year, or who have traveled more than three time zones during the one month prior to the study will be excluded.
* Pregnant women, decisionally impaired adults, and prisoners will be excluded.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Vascular Endothelial Function | 2 weeks
  Investigators will measure endothelial function as flow-mediated dilation.
Cardiovascular Risk | 2 weeks
  Investigators will measure cardiovascular risk as carotid intima-media thickness (IMT).
Coronary Atherosclerotic Burden | 2 weeks
  Investigators may measure coronary atherosclerotic measure from a computerized tomography (CT) scan. This measure is optional for participants.
  The scan will be used to calculate coronary artery calcium score (CAC score and/or Agatston score). The CAC score indicates risk of future coronary artery events. A CAC score of 0 indicates absence of coronary artery calcification. A score of 0 is very low risk, and risk increases with increasing numbers (e.g. 100-300 is increased risk, >300 is very high risk). Higher scores may indicate higher risk of future coronary events.
  The Agatston score is also an atherosclerotic measure that may indicate risk of future coronary artery events. Agatston also goes up from 1 on a linear scale (e.g. 1-100 is discreet atherosclerosis, up to 400 is moderate, >400 is severe).
Heart rate | 2 weeks
  Heart rate will be measured as beats per minute while participants are in a supine position.
Blood pressure | 2 weeks
  Blood pressure (systolic and diastolic) will be measured in a supine position in the dominant arm.
24-hour BP measurement | 2 weeks
  Investigators will measure 24-hour ambulatory blood pressure (AMBP, Spacelabs, Inc) for 24-h period before each in-lab visit, including the optional visit. Both systolic and diastolic blood pressure will be measured.
Sleep duration | 2 weeks
  Sleep duration will be scored from the ActiGraph and correlated with the sleep and activity diary.
Sleep efficiency | 2 weeks
  Sleep efficiency will be scored from the ActiGraph and correlated with the sleep and activity diary. Sleep efficiency measures amount of time asleep while in bed. This is measured from 0-100%, where 0 indicates low sleep efficiency, or no sleep in bed, and higher percent indicates more sleep, or higher sleep efficiency while in bed.
Physical Activity | 2 weeks
  Activity will be scored from the ActiGraph and correlated with the sleep and activity diary.
Total Mood Disturbance | 2 weeks
  Total Mood Disturbance will be measured from the Profile of Mood States (POMS) questionnaire. Participants will rate their mood states on a likert scale of 0-4. POMS may indicate both positive and negative moods. There is a minimum score of 0, and maximum of 260. In general, lower scores indicate less mood disturbance, while higher scores indicate higher mood disturbance. Subsets of particular scores may indicate particular mood states.
Timing of caloric intake | 2 weeks
  Timing of caloric intake may be measured by participant completion of a 7-day photographic food diary before the in-lab visits. MealLoggerTM(Wellness Foundry, New York, http://www.meallogger.com). Photographs are time stamped, indicating timing of caloric intake.
Content of caloric intake | 2 weeks
  Content of caloric intake may be measured by participant completion of a 7-day photographic food diary before the in-lab visits. MealLoggerTM(Wellness Foundry, New York, http://www.meallogger.com) These photographs may be assessed to identify micronutrients and macronutrients in content of food.
Blood Cholesterol | 2 weeks
  Blood cholesterol (measured in plasma according to laboratory values) may be measured by a complete blood count after blood draw. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
Blood fasting glucose | 2 weeks
  Blood fasting glucose (measured in plasma according to laboratory values) may be measured by a complete blood count after blood draw. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
C-reactive protein | 2 weeks
  C-reactive protein (measured in plasma according to laboratory values) may be measured by lab tests after blood draw as a blood inflammatory marker. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
Interleukins | 2 weeks
  Interleukin 6 (IL-6), Interleukin 1(IL-1 β), interleukin-1 receptor antagonist (IL-1RA), interleukin 18 (IL-18), measured in plasma according to laboratory values, may be measured by lab tests after blood draw as blood inflammatory markers. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
Plasminogen activator inhibitor-1 | 2 weeks
  Plasminogen activator inhibitor-1 (measured in plasma according to laboratory values) may be measured by lab tests after blood draw as a blood inflammatory marker. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
P-selectin | 2 weeks
  P-selectin (measured in plasma according to laboratory values) may be measured by lab tests after blood draw as a blood inflammatory marker. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
Blood cortisol | 2 weeks
  Cortisol (measured in plasma according to laboratory values) may be measured by lab tests after blood draw as a measure of stress. This is a hypothesis generating variable. Higher values may indicate increased cardiovascular risk.
Body Mass Index (BMI) | 2 weeks
  Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh S Thosar, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No